CLINICAL TRIAL: NCT05243095
Title: The Effect of Computer-Assisted, Game-Based Cognitive Training on Attention: A Randomized Controlled Study
Brief Title: Computer-Assisted, Game-Based Cognitive Training on Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Ünal, PT.,PhD., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27.01.2022/Attention
Record Dates: First submitted 2022-01-27; First posted 2022-02-16 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Young Adults; Attention
Keywords: Cognitive-training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training group (Experimental): The training group received 20 minutes of cognitive training every day for 8 weeks
  Interventions: Other: Computer assited, game-based cognitive training
- Control group (No Intervention): No training was applied to the control group.

INTERVENTIONS:
Other: Computer assited, game-based cognitive training — After recording the demographic information of the participants, the Stroop Test was applied to evaluate attention. After the stages of the test were explained to the participants in detail, they were shown once in practice.
  The training group received 20 minutes of cognitive training every day for 8 weeks. No training was applied to the control group. Groups were evaluated at baseline and after 8 weeks.
  Arms: Cognitive training group

SUMMARY:
The aim of this study was to investigate the effect of 8 weeks of cognitive training on attention function in healthy young people.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 21-24,
* No communication problem,
* Not continuing any exercise program for the last 1 year,
* Having a smart phone, tablet or computer required to participate in the training program,
* Individuals who volunteered to participate in the study.

Exclusion Criteria:

* Having vision and hearing problems,
* Individuals who continued the physical exercise program and/or had hobbies such as puzzles and jigsaw puzzles that could affect the cognitive level.

Ages: 21 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Stroop test | 10 minutes
  The Stroop Test is a test that evaluates frontal lobe functions and cognitive processes such as attention and information processing.
  The Stroop Test TBAG Form consists of four white cards measuring 14.0 x 21.5 cm.
  The performance of the participants was scored according to three separate criteria for each section: These criteria are: the time taken until the last item of the section is answered with the "start" command, the number of errors, the number of corrected responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No